CLINICAL TRIAL: NCT01461603
Title: Local Effects of Amino Acids and 3-hydroxybutyrate in the Bilaterally Perfused Human Leg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-20110177
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-01

CONDITIONS: Critical Illness; Protein Metabolism; Pharmaconutrients
Keywords: critical illness; protein metabolism; pharmaconutrients
MeSH Terms: conditions — Critical Illness | interventions — amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amino acids (Active Comparator): Amino acids compared to saline
  Interventions: Dietary Supplement: Vamin (Fresenius Kabi)
- 3hydroxybutyrat (3OHB) (Active Comparator): Ketone body, 3OHB compared to saline
  Interventions: Dietary Supplement: 3hydroxybutyrate

INTERVENTIONS:
Dietary Supplement: Vamin (Fresenius Kabi) — Vamin 18gN 1ml/min infusion in 6 hours
  Arms: Amino acids
Dietary Supplement: 3hydroxybutyrate — Goldbio, FFA-3OHB, dry powder mixed with sterile water at Aarhus University hospital pharmacy.
  Other Names: 3OHB, 3hydroxybutyric acid
  Arms: 3hydroxybutyrat (3OHB)

SUMMARY:
Introduction: Protein loss during critical illness is an important problem and is shown to predict overall survival. In animal studies, infusion of leucine is shown to increase the synthesis of muscle protein by 30-40% and decrease protein degradation by 30%.

Objectives: Compared to saline, an amino acid or 3hydroxybutyrate infusion in the femoral artery will promote protein synthesis and inhibit breakdown assessed with local a/v phenylalanine and tyrosine tracer kinetics in healthy volunteers. These effects will include distinct alterations in muscle signal events, in particular mTOR.

Methods: n = 10 healthy male subjects are equipped with catheters in aa. femorals and vv. femorals bilaterally under local anaesthetics. Each study comprises a 3-hour basal period and a 3-hour period with hyperinsulinaemic-euglycaemic clamp. During the test, samples of arterial and venous blood and 4 muscle biopsies are obtained. The intervention contain continues saline infusion compared to either amino acids (Vamin) or 3hydroxybutyrate solution FFa-3OHB.

Perspectives: This study elucidates the direct effect of aminoacids and ketone bodies on muscle protein metabolism in humans and contribute to further development of nutritional therapy in human catabolic states.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 28
* Written consent before study start

Exclusion Criteria:

* Diabetes
* Inclusion in other studies using ionizing radiation.
* Allergic to egg or soy

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle metabolism after administration of amino acids. | Basal period and a glucose clamp (6 hours pr.day)
  Measured by arterio-venous differences of isotope tracers

SECONDARY OUTCOMES:
Intracellular mTOR and pAkt signal activation after infusion of amino acids. | Basal period and a glucose clamp (6 hours pr. day)
  4 muscle biopsies measured for mTOR and pAkt activation by western blotting

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Dr.Med., Principal Investigator — University of Aarhus
Locations (1):
- M-researchlab. MEA, Aarhus University Hospital, NBG, Aarhus C, Denmark